CLINICAL TRIAL: NCT00760279
Title: An Open Label Evaluation of the Pharmacokinetics and Safety of Single Dose Intravenous Azithromycin in Preterm Neonates Pediatric Pharmacology Research Unit, Children's Hospital of Michigan
Brief Title: An Open Label Evaluation of the Pharmacokinetics and Safety of Single Dose Intravenous Azithromycin in Preterm Neonates
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD) (NIH)
Collaborators: Pediatric Pharmacology Research Units Network (Network); Children's Hospital of Michigan (Other)
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: PPRU10820
Record Dates: First submitted 2008-09-25; First posted 2008-09-26 (Estimated); Last update posted 2008-09-26 (Estimated); Status verified 2008-09

CONDITIONS: Ureaplasma; Bacterial Infection
Keywords: Bacterial infection; Azithromycin
MeSH Terms: conditions — Bacterial Infections | interventions — Azithromycin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Drug: Azithromycin

SUMMARY:
The purpose of this study is to evaluate the pharmacokinetics and safety of a single dose of IV azithromycin in preterm neonates and confirm that the pharmacokinetics of azithromycin is similar in the 24-<32 week and 32-<37 week neonate. The dose of 10 mg/kg has been chosen on the basis of previous pediatric pharmacokinetic studies.

DETAILED DESCRIPTION:
In vitro studies with azithromycin show good inhibitory activity against U. urealyticum. Pharmacokinetic studies of azithromycin in older children show better tolerance, higher tissue concentration, fewer side effects, and fewer drug interactions, when compared to erythromycin. Thus far, there have been no published data on the pharmacokinetic profile of azithromycin in neonates including low birth weight infants. However, the clinical pharmacology profile suggests a substantial therapeutic advantage of this drug in the newborn. To date, there are no data on the PK profile of IV Azithromycin from whence rational dosing can be derived.

ELIGIBILITY:
Inclusion Criteria:

1. 24 to 37 weeks gestational age
2. postnatal age 0 to 30 days
3. May require therapy with antibiotics/anti-infectives
4. Have baseline Hematology labs available (hemoglobin, hematocrit, white blood cell and differential and platelet count), which have been obtained within the previous 72 hours, as part of their standard of care
5. Signed informed consent by the parent or guardian

Exclusion Criteria:

1. Clinically significant hepatic disease (ALT or AST twice the normal value)
2. Clinically significant anemia (hemoglobin < 10 gm %)
3. Neutropenia (absolute neutrophil count < 500 cells/mm3)
4. Clinically significant renal disease [Creatinine clearance twice the normal value, as calculated by the Schwartz formula : Length in cms x k (a constant) / S.Cr (Values for the constant are given in Appendix 1)]
5. Cardiac rhythm abnormalities
6. Critically ill patients
7. Patients who are on or expected to be on the following concurrent medications carbamazepine, phenytoin, theophylline, digoxin, warfarin, ergot alkaloids, triazolam, cyclosporine, terfenadine, hexobarbital and antacids.

Max Age: 30 Days | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 16 (Estimated)
Dates: Start 2005-09

PRIMARY OUTCOMES:
Safety: Patients will be monitored for clinical adverse events and have standard hematology labs drawn within 72 hours of study entry. Liver function tests, renal function tests and standard chemistries will be drawn prior to and at the end of the study.

CONTACTS AND LOCATIONS:
Overall Officials: Elias Tessema, M.D., Principal Investigator — Wayne State; David Edwards, Pharm.D., Principal Investigator — Wayne State; Jacob Aranda, M.D., Ph.D., Principal Investigator — Wayne State
Locations (2):
- United States (2):
  - Wayne State, Detroit, Michigan
  - Rainbow Babies and Children's Hospital, Cleveland, Ohio